CLINICAL TRIAL: NCT05527379
Title: Interest of Virtual Reality to Reduce Patient Anxiety During the Placement of a Percutaneous Implantable Port Catheter
Acronym: RV-CIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0824
Record Dates: First submitted 2022-08-24; First posted 2022-09-02 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Anxiety; CIP
Keywords: virtual reality; anxiety; CIP
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CIP procedure under virtual reality (Experimental): CIP procedure under virtual reality
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — When the patient is ready to have the CIP procedure the tablet will be presented to him so that he can view and choose the immersive film that suits him best.
  Before fitting the virtual reality helmet and the start of the film, the patient's anxiety will be evaluated by ENS on a scale of 0 to 10 . The patient's anxiety will also be evaluated at the end of the procedure.
  The patient will be contacted by telephone by an investigator between D+1 and D+5 in order to reassess and remotely from the pose, his memorization of the gesture and to look for adverse events.

SUMMARY:
The Vascular Access Unit (UAV) of the Lyon Sud Hospital Center is the first unit within a French public establishment where the Regional Health Agency (ARS) has authorized that medical procedures for the installation of central venous access be performed by nurses.

The installation of CIP represents an anxiety-provoking step for the patient, because the gesture, which consists of inserting a box under the skin, connected to a catheter, placed in a deep vein, involves uncomfortable, even painful moments. In the UAV, the installation of this device is carried out in the operating room, without premedication and only under local anesthesia. Affected patients usually have a diagnosis of serious illness (oncology).

Virtual Reality (VR) simulates the physical presence of the patient in an environment artificially generated by software. Many applications have already been evaluated in different health sectors, the investigators would like to show its interest in reducing patient anxiety during CIP placement under local anesthesia, without premedication.

The medical device used is Lumeen. It is a Class I medical device software within the meaning of Regulation (EU) 2017/745, CE marked. In the context of research, the Relaxation module is used. This module is the one intended for the management of anxiety and pain induced by medical procedures in adults and children over 6 years of age. It allows to perform immersions in 360° videos in real shots or computer-generated images, accompanied by natural sounds, relaxing music and a relaxation script recorded by hypnotherapists. The duration of an immersion can be adjusted according to the needs of the medical procedure..

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥18 years old
* Patient operated on an outpatient basis and available for a phone call between D+1 and D+5
* Patient operated for a 1st pose of CIP at the UAV
* Patient whose anxiety measured by ENS Anxiety is at least 4/10 at entry
* Patient having signed the Informed Consent
* Patient affiliated to a social security

Exclusion Criteria:

* Patient not sufficiently fluent in the French language, in the judgment of the investigator, to allow him a good understanding of the implementation and the interest of the virtual reality headset material;
* Patient with motion sickness;
* Patient participating in another study who, in the judgment of the investigator, could interfere with the results of this research protocol;
* Patient deprived of liberty or placed under guardianship or curators;
* Pregnant or breastfeeding women;
* Patient with a history of epilepsy ;
* Patient with a pacemaker or pacemaker;
* Patient with psychiatric disorders of a psychotic nature in the acute phase or visual hallucinations;
* Patient under anxiolytic treatment;
* Patient presenting wounds or infections on the level of the head not allowing the installation of the virtual reality helmet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Description of Patient's anxiety through his participation | through study completion, an average of 5 days
  Evaluated by Simple Numerical Scale : Anxiety from 0 to 10
Evolution of Patient's anxiety during the procedure | Day 0
  Evaluated by Simple Numerical Scale : Anxiety from 0 to 10

SECONDARY OUTCOMES:
Effects of virtual reality on the pain perceived by the patient; | Day 0 (after placing the port)
  The patient's pain, over the entire procedure, measured by Simple Numerical Scale : Pain from 0 to 10
Effects of virtual reality on Pulse | Day 0 (before, during and after placing the port)
  The Pulse of the patient
Effects of virtual reality on Blood Pressure | Day 0 (before, during and after placing the port)
  The Blood Pressure of the patient (both systolic and diastolic)
Effects of virtual reality on memorization of the gesture | Day 0 (after placing the port) and through study completion between D+1 and D+5
  Measured by a Likert scale (Likert scale = Very Uncomfortable- Uncomfortable- Comfortable- Very Comfortable)
Effects of virtual reality on the perception of time | Day 0 (after placing the port)
  Perception of time in minutes estimated by the patient (In your opinion, how long did the gesture last? and difference with the actual duration of the gesture
Effects of virtual reality on satisfaction and comfort during installation | Day 0 (after placing the port)
  Measured by a Simple Numerical Scale from 0 to 10
Effects of virtual reality on the caregiver's perception of the ease of the gesture | Day 0 (after placing the port)
  Measured by a Likert scale, (Likert scale = Easy-patient Immobile - appearing relaxed / Moderately Easy-Patient slightly mobile- Reactive / Difficult-Patient having difficulty in staying Still- Very reactive- Seeming tense)
Effects of virtual reality on caregiver satisfaction | Day 0 (after placing the port)
  Measured by a Simple Numerical Scale from 0 to 10
Effects of virtual reality on the duration of the intervention | Day 0 (after placing the port)
  Duration of the procedure in minutes between the patient entering and leaving the operating room

CONTACTS AND LOCATIONS:
Overall Officials: Annie de FILIPPIS, Principal Investigator — HCL
Locations (1):
- Unité d'Accès Vasculaire/Secteur Anesthésie Blocs - CHLS, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No